CLINICAL TRIAL: NCT02102204
Title: A Multicenter Single-arm Extension Study to Describe the Long-term Safety of AMG 416 in the Treatment of Secondary Hyperparathyroidism in Subjects With Chronic Kidney Disease on Hemodialysis
Brief Title: Extension Study of Etelcalcetide for Treatment of Secondary Hyperparathyroidism in Patients With Chronic Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130213; 2013-004136-30 (EudraCT Number); KAI-4169 (Other: KAI Pharmaceuticals (wholly owned subsidiary of Amgen, Inc.))
Record Dates: First submitted 2014-03-03; First posted 2014-04-02 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperparathyroidism (SHPT), chrominc kidney disease (CKD), hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Etelcalcetide (Experimental): Participants received etelcalcetide three times a week (TIW) by bolus injection at the end of hemodialysis. The minimum etelcalcetide dose in this study was 2.5 mg and the maximum dose was 15 mg. Etelcalcetide dose was titrated to maintain parathyroid hormone levels within 2x to 9x the upper limit of normal based on the reference range of the assay used at the individual study center.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Etelcalcetide was supplied as a sterile, preservative-free, ready-to-administer aqueous solution.
  Other Names: KAI-4169; AMG 416; Parasabiv

SUMMARY:
This is a multicenter, single-arm, extension study to characterize the long-term safety and tolerability of etelcalcetide in the treatment of Secondary Hyperparathyroidism (SHPT) in adults with Chronic Kidney Disease (CKD) on hemodialysis.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, extension study in which adults with secondary hyperparathyroidism currently receiving hemodialysis and previously treated in Amgen studies 20120231 (NCT01785875), 20120334 (NCT01576146), or 20120360 (NCT01896232) will continue to be treated with etelcalcetide until approximately 2.5 years after the first participant was enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Subject has completed treatment in Study 20120231 (also known as KAI-4169-008) or Study 20120360, or has participated in Study 20120334 (also known as KAI-4169-005-01)
* Female subjects who are: post-menopausal (post-menopausal is defined as no menses for the previous 1 year and over the age of 50 years), surgically sterilized, have a medical condition that prevents pregnancy, remain abstinent, or are willing to use an acceptable method of effective contraception during the study and for 3 months after the last dose. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 2 weeks prior to the first dose of AMG 416 in the current study
* Subject must be receiving hemodialysis 3 or 4 times weekly for at least 3 months

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study (other than in one of the designated parent studies)
* Subject has known sensitivity to any of the products or components to be administered during dosing
* Subject has been prescribed cinacalcet by the primary nephrologist between the conclusion of the parent study and the start of dosing with AMG 416 in the current study
* Subject is receiving dialysis prescription dialysate calcium concentration < 2.25 mEq/L
* Subject is pregnant or nursing

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (205):
- United States (67):
  - Research Site, Birmingham, Alabama
  - Research Site, Alhambra, California
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Cudahy, California
  - Research Site, Granada Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Simi Valley, California
  - Research Site, Vacaville, California
  - Research Site, Whittier, California
  - Research Site, Aurora, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Dublin, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Highland Park, Illinois
  - Research Site, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Brookhaven, Mississippi
  - Research Site, Columbus, Mississippi
  - Research Site, Gulfport, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Eatontown, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, College Point, New York
  - Research Site, Great Neck, New York
  - Research Site, Mineola, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Yonkers, New York
  - Research Site, Durham, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Fairfax, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Mechanicsville, Virginia
  - Research Site, Bluefield, West Virginia
- Australia (6):
  - Research Site, Liverpool, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Prahan, Victoria
- Austria (4):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Baudour
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Hasselt
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
  - Research Site, Tournai
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Brampton, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Czechia (7):
  - Research Site, Hradec Králové
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Slavkov u Brna
  - Research Site, Ústí nad Orlicí
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Fredericia
- France (8):
  - Research Site, Caen
  - Research Site, La Tronche
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Reims
  - Research Site, Saint-Ouen
  - Research Site, Saint-Priest-en-Jarez
- Germany (9):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Langenhagen
  - Research Site, Minden
  - Research Site, München
  - Research Site, Villingen-Schwenningen
  - Research Site, Wiesbaden
  - Research Site, Zwickau
- Greece (5):
  - Research Site, Alexandroupoli
  - Research Site, Larissa
  - Research Site, Nikaia, Piraeus
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (11):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Szigetvár
  - Research Site, Zalaegerszeg
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (10):
  - Research Site, Ancona
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Lucca
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Pordenone
  - Research Site, Verona
- Research Site, Riga, Latvia
- Lithuania (3):
  - Research Site, Alytus
  - Research Site, Kaunas
  - Research Site, Ukmerge
- Netherlands (2):
  - Research Site, Rotterdam
  - Research Site, Venlo
- Research Site, Hamilton, New Zealand
- Poland (12):
  - Research Site, Gdansk
  - Research Site, Golub-Dobrzyń
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Sieradz
  - Research Site, Wadowice
  - Research Site, Warsaw
  - Research Site, Zabrze
  - Research Site, Zamość
  - Research Site, Żyrardów
- Portugal (8):
  - Research Site, Almada
  - Research Site, Aveiro
  - Research Site, Forte Da Casa
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Santo Tirso
  - Research Site, Setúbal
  - Research Site, Vila Franca de Xira
- Russia (5):
  - Research Site, Mitishi
  - Research Site, Moscow
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Spain (10):
  - Research Site, Córdoba, Andalusia
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Badajoz, Extremadura
  - Research Site, Majadahonda, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Torrevieja, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (4):
  - Research Site, Karlstad
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Uppsala
- Switzerland (6):
  - Research Site, Aarau
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Locarno
  - Research Site, Zurich
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 229 study centers in Europe, Australia, New Zealand, and North America
Pre-assignment Details: A total of 902 participants were enrolled in Study 20130213: 215 and 200 participants from the cinacalcet and etelcalcetide groups of the double-blind parent Study 20120360 (NCT01896232), respectively, and 487 participants from the open-label parent Studies 20120231 (NCT01785875) and 20120334 (NCT01576146).
Period: Overall Study
Arm/Group | Etelcalcetide
Started | 902
Received Etelcalcetide | 884
Completed | 598
Not Completed | 304
Not completed — Withdrawal by Subject | 137
Not completed — Death | 92
Not completed — Lost to Follow-up | 65
Not completed — Sponsor Decision | 5
Not completed — Ongoing | 5

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all participants who received at least 1 dose of etelcalcetide in the current study (20130213).
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 884
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 582
  ≥ 65 years | 302
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357
  Male | 527
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 78
  Not Hispanic or Latino | 806
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 14
  Black | 192
  Native Hawaiian or Other Pacific Islander | 9
  White | 657
  Other | 11
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] — Starting values are presented in this table, and are defined as the first non-missing measurement within the first 3 months on or after analysis day 1 (inclusive). Population: Participants with non-missing data
  pg/mL
    number analyzed (Participants) | 855
    (all) | 528.3 (566.4)
Albumin Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] — Starting values are presented in this table, and are defined as the first non-missing measurement within the first 3 months on or after analysis day 1 (inclusive). Population: Participants with non-missing data
  mg/dL
    number analyzed (Participants) | 875
    (all) | 8.94 (0.79)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Starting values are presented in this table, and are defined as the first non-missing measurement within the first 3 months on or after analysis day 1 (inclusive). Population: Participants with non-missing data
  mg/dL
    number analyzed (Participants) | 875
    (all) | 5.24 (1.69)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event is an AE that met at least 1 of the following criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
  The relationship of each AE to study treatment was assessed by the investigator.
  The following AE grading scale was used:
  Mild: Transient or mild discomfort; no limitation in activity; no medical intervention/therapy required Moderate: Mild to moderate limitation in activity-some assistance may be needed; no or minimal medical intervention/therapy required Severe: Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalization possible Life-threatening: Extreme limitation in activity, significant assistance required, significant medical intervention/therapy required, hospitalization probable.
Time Frame: From the date of first dose of etelcalcetide (in the current study) and up to 30 days after the last dose; median duration of treatment was 563 days.
Population: Participants who received at least 1 dose of etelcalcetide in the current study (20130213).
Measure: Number; unit: participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 884
participants
  Any adverse event | 768
  Serious adverse events | 436
  Treatment-related adverse events | 287
  Serious treatment-related adverse events | 4
  AEs leading to discontinuation of etelcalcetide | 41
  Fatal adverse events | 89
  Mild adverse events | 123
  Moderate adverse events | 219
  Severe adverse events | 324
  Life-threatening adverse events | 102

2. Secondary Outcome: Percentage of Participants With Parathyroid Hormone Levels Between Two to Nine-times the Upper Limit of Normal
Description: The percentage of participants who maintained plasma parathyroid hormone (PTH) levels within the Kidney Disease Improving Global Outcomes (KDIGO) recommended range of not less than 2x the upper limit of normal (ULN) and not greater than 9x the ULN at months 6, 12, and 18, with the ULN based on the reference range of the assay used at the individual clinical site.
Time Frame: Months 6, 12, and 18
Population: Participants who received at least 1 dose of etelcalcetide in the current study (20130213) with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 884
percentage of participants
  Month 6: number analyzed (Participants) | 770
  Month 6 | 67.0 [63.6 to 70.3]
  Month 12: number analyzed (Participants) | 679
  Month 12 | 73.2 [69.7 to 76.5]
  Month 18: number analyzed (Participants) | 540
  Month 18 | 71.9 [67.9 to 75.6]

3. Secondary Outcome: Percentage of Participants With Serum Phosphorus ≤ the ULN
Description: Percentage of participants with serum phosphorus less than or equal to the upper limit of normal for the assay used.
Time Frame: Months 6, 12, and 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 884
percentage of participants
  Month 6: number analyzed (Participants) | 744
  Month 6 | 39.4 [35.9 to 43.0]
  Month 12: number analyzed (Participants) | 625
  Month 12 | 40.0 [36.1 to 44.0]
  Month 18: number analyzed (Participants) | 478
  Month 18 | 36.8 [32.5 to 41.3]

4. Secondary Outcome: Percentage of Participants With Serum Corrected Calcium < 7.5 mg/dL
Description: The percentage of participants with serum corrected calcium (cCa) reported for cumulative time intervals from day 1 through months 6, 12, and 18, using the participant's lowest recorded corrected calcium value during the time interval.
  If serum albumin was less than 4.0 g/dL, serum calcium was corrected according to the following formula:
  cCa (mg/dL) = total calcium (mg/dL) + (4 - albumin [g/dL])*0.8. If serum albumin was > 4.0 g/dL no correction was made.
Time Frame: From day 1 to months 6, 12, and 18
Population: Participants who received at least 1 dose of etelcalcetide in the current study (20130213) with available data at the beginning of the time interval.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 871
percentage of participants
  Day 1 to Month 6 | 9.5 [7.7 to 11.7]
  Day 1 to Month 12 | 14.1 [11.9 to 16.6]
  Day 1 to Month 18 | 16.3 [13.9 to 18.9]

5. Secondary Outcome: Number of Participants With Shifts From Baseline Grade 0 or 1 to Postbaseline Grade 3 or 4 for Laboratory Parameters
Description: The Common Terminology Criteria for Adverse Events (CTCAE) grades for laboratory parameter values were defined based on the upper/lower limit of normal from the local laboratories contracted by the study centers.
Time Frame: Baseline to end of treatment; median duration of treatment was 563 days.
Population: Participants who received at least 1 dose of etelcalcetide in the current study (20130213).
Measure: Number; unit: participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 884
participants
  Increased Alanine Aminotransferase Grade 1 to 3 | 1
  Increased Alkaline Phosphatase Grade 1 to 3 | 2
  Increased Aspartate Aminotransferase Grade 1 to 3 | 1
  Decreased Corrected Calcium Grade 1 to 3 | 18
  Decreased Corrected Calcium Grade 1 to 4 | 2
  Decreased ionized Calcium Grade 1 to 3 | 1
  Decreased ionized Calcium Grade 1 to 4 | 2
  Decreased Phosphorous Grade 1 to 3 | 1

6. Secondary Outcome: Number of Participants Who Developed Positive Binding Anti-Etelcalcetide Antibodies
Description: The number of participants who were binding antibody positive post-baseline with a negative or no result at baseline (where baseline for participants previously treated with etelcalcetide is Day 1 of the first study in which they were exposed to etelcalcetide and for participants previously treated with cinacalcet is the ending time point for study 20120360).
Time Frame: Baseline and every 6 months (up to 24 months)
Population: Participants who received at least 1 dose of etelcalcetide in the current study with a post-baseline antibody result during this study
Measure: Number; unit: participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 808
participants | 111

ADVERSE EVENTS:
Time Frame: From the date of first dose of etelcalcetide (in the current study) and up to 30 days after the last dose; median duration of treatment was 563 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 436/884
Other Adverse Events (participants affected / at risk) | 519/884
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=884)
Anaemia (Blood and lymphatic system disorders) | 19
Coagulopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 13
Angina pectoris (Cardiac disorders) | 8
Angina unstable (Cardiac disorders) | 4
Aortic valve incompetence (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 15
Atrial flutter (Cardiac disorders) | 3
Atrioventricular block complete (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 20
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 8
Cardiac valve disease (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 4
Cardiogenic shock (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 7
Coronary artery stenosis (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 7
Myocardial ischaemia (Cardiac disorders) | 5
Pericardial effusion (Cardiac disorders) | 2
Pericarditis uraemic (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 3
Ventricular tachycardia (Cardiac disorders) | 2
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 4
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Porencephaly (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Goitre (Endocrine disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 1
Cataract (Eye disorders) | 2
Optic ischaemic neuropathy (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 3
Colitis ischaemic (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastroduodenitis (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 3
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Hernial eventration (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal ischaemia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 2
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatic disorder (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 4
Pancreatitis acute (Gastrointestinal disorders) | 5
Pancreatitis chronic (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestine polyp (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 5
Chest pain (General disorders) | 7
Death (General disorders) | 4
Drowning (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 3
Hyperpyrexia (General disorders) | 1
Impaired healing (General disorders) | 2
Ischaemic ulcer (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 11
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 11
Sudden death (General disorders) | 4
Systemic inflammatory response syndrome (General disorders) | 2
Acute hepatic failure (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 3
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 7
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Gallbladder disorder (Hepatobiliary disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic cyst ruptured (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1
Chronic allograft nephropathy (Immune system disorders) | 1
Transplant rejection (Immune system disorders) | 2
Abdominal abscess (Infections and infestations) | 1
Abdominal wall abscess (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Arteriovenous fistula site infection (Infections and infestations) | 3
Arteriovenous graft site abscess (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 3
Arthritis bacterial (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 3
Bacterial sepsis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 10
Bronchitis bacterial (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 9
Cellulitis gangrenous (Infections and infestations) | 1
Cellulitis orbital (Infections and infestations) | 1
Citrobacter sepsis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 7
Device related sepsis (Infections and infestations) | 4
Diabetic foot infection (Infections and infestations) | 2
Diabetic gangrene (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 7
Epiglottitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 2
Febrile infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 9
Gastroenteritis (Infections and infestations) | 7
Helicobacter gastritis (Infections and infestations) | 1
Hepatitis A (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Intervertebral discitis (Infections and infestations) | 3
Intestinal tuberculosis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Localised infection (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 4
Lower respiratory tract infection viral (Infections and infestations) | 1
Mediastinitis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 11
Osteomyelitis chronic (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 40
Post procedural infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 7
Respiratory tract infection viral (Infections and infestations) | 3
Sepsis (Infections and infestations) | 27
Septic shock (Infections and infestations) | 14
Serratia bacteraemia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 3
Staphylococcal sepsis (Infections and infestations) | 1
Stoma site infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 2
Systemic infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 6
Urosepsis (Infections and infestations) | 3
Vascular access site infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Vulval abscess (Infections and infestations) | 1
Wound infection (Infections and infestations) | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 24
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 9
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 7
Femur fracture (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 3
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Shunt aneurysm (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 2
Shunt stenosis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 5
Vascular access malfunction (Injury, poisoning and procedural complications) | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Vascular injury (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Blood potassium decreased (Investigations) | 1
Paracentesis (Investigations) | 1
Peripheral pulse decreased (Investigations) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 16
Fluid retention (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 16
Hypervolaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 2
Brain stem stroke (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 4
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 5
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 7
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 3
Epilepsy (Nervous system disorders) | 2
Facial paresis (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Metabolic encephalopathy (Nervous system disorders) | 3
Multiple sclerosis (Nervous system disorders) | 1
Neuritis cranial (Nervous system disorders) | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Quadriplegia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 13
Transient global amnesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 1
Uraemic neuropathy (Nervous system disorders) | 1
Device dislocation (Product Issues) | 2
Device failure (Product Issues) | 1
Device malfunction (Product Issues) | 1
Device occlusion (Product Issues) | 1
Stent malfunction (Product Issues) | 1
Thrombosis in device (Product Issues) | 6
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Depression suicidal (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 8
Suicide attempt (Psychiatric disorders) | 1
End stage renal disease (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 2
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal vein thrombosis (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Priapism (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dependence on respirator (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Diabetic foot (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Accelerated hypertension (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Exsanguination (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 3
Haematoma (Vascular disorders) | 4
Hypertension (Vascular disorders) | 9
Hypertensive crisis (Vascular disorders) | 6
Hypertensive emergency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 8
Hypovolaemic shock (Vascular disorders) | 1
Iliac artery occlusion (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 3
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 7
Peripheral vascular disorder (Vascular disorders) | 4
Shock haemorrhagic (Vascular disorders) | 1
Steal syndrome (Vascular disorders) | 2
Superior vena cava stenosis (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 2
Thrombophlebitis (Vascular disorders) | 1
Vascular calcification (Vascular disorders) | 1
Vascular compression (Vascular disorders) | 1
Venous occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=884)
Diarrhoea (Gastrointestinal disorders) | 84
Nausea (Gastrointestinal disorders) | 58
Vomiting (Gastrointestinal disorders) | 55
Upper respiratory tract infection (Infections and infestations) | 58
Blood calcium decreased (Investigations) | 251
Hyperphosphataemia (Metabolism and nutrition disorders) | 81
Back pain (Musculoskeletal and connective tissue disorders) | 51
Muscle spasms (Musculoskeletal and connective tissue disorders) | 73
Pain in extremity (Musculoskeletal and connective tissue disorders) | 59
Cough (Respiratory, thoracic and mediastinal disorders) | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49
Hypertension (Vascular disorders) | 62
Hypotension (Vascular disorders) | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.